CLINICAL TRIAL: NCT05613920
Title: Dietary Management of Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Wenyao Geng, Principal Investigator, Qingdao University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: QDU-HEC-2021149
Record Dates: First submitted 2022-10-21; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Diet; Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diet management program based on the nudge strategy (Experimental): The intervention group will receive a diet management program based on the nudge strategy
  Interventions: Behavioral: diet management program based on the nudge strategy
- routine dietary management program (No Intervention): The control group will receive a routine dietary management program

INTERVENTIONS:
Behavioral: diet management program based on the nudge strategy — The intervention group received a 12-week dietary management intervention based on the nudge strategy. The MINDSPACE framework was used, which has nine intervention categories. Face-to-face intervention and telephone follow-up were used to provide targeted dietary management.
  Arms: diet management program based on the nudge strategy

SUMMARY:
The goal of this clinical trial is to test effect of dietary management program based on the nudge strategy in gestational diabetes mellitus patients. The main questions it aims to answer is whether the dietary management program is effective for the diet management behavior of gestational diabetes mellitus patients.

Participants will receive a 12 week dietary management program. The intervention group will receive a diet management program based on the nudge strategy, and the control group will receive a routine dietary management program. Researchers will compare two group's glycemic control and pregnancy outcomes and to see if effective for the diet management behavior.

ELIGIBILITY:
Inclusion criteria

1. Meeting the diagnostic criteria related to GDM by oral glucose tolerance test (OGTT), etc.
2. Singleton pregnancy
3. Age ≥ 18 years
4. Gestational weeks 24-28
5. Informed consent for voluntary participation in this study Exclusion criteria

1.Patients with significant heart, liver, lung and other organ failure and malignancy 2.Previous history of psychiatric disorders or existing psychiatric disorders 3.Diabetes combined with other complications such as gestational hypertension Dropout criteria

1. Lost to the study due to unforeseen circumstances
2. Voluntarily requested to withdraw from the study
3. Did not take the intervention as required by the relevant requirements
4. Condition was unstable and could not continue to cooperate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Changes in blood glucose levels over time | Pre-intervention, 1-month post-intervention and 3-months post-intervention
  With the change of intervention and time, it is better for the fasting blood glucose to decrease; With the change of intervention and time, it is better that the 1hPG decreases; With the change of intervention and time, it is better that the 2hPG decreases.

SECONDARY OUTCOMES:
pregnancy outcomes | During the delivery of pregnant women, the relevant data of pregnancy outcome were collected by consulting medical records or telephone follow-up.
  Number of Participants with Premature, Cesarean delivery, Gestational hypertension, Giant baby, Fetal intrauterine distress

OTHER OUTCOMES:
Apgar score of newborn | Apgar score at 1 minute and 5 minutes after birth
  Apgar score at 1 minute and 5 minutes after birth in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Wenyao Geng, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Decide not to share participant data from the perspective of protecting participant privacy

REFERENCES:
- [Result] Phillips JK, Skelly JM, Roberts LM, Bernstein IM, Higgins ST. Combined financial incentives and behavioral weight management to enhance adherence with gestational weight gain guidelines: a randomized controlled trial. Am J Obstet Gynecol MFM. 2019 Mar;1(1):42-49. doi: 10.1016/j.ajogmf.2019.02.002. Epub 2019 Mar 5. PMID 33319756
- [Result] Xu S, Yu Q, Mi J, Li H. Clinical efficacy of nutritional diet therapy on gestational diabetes mellitus. Am J Transl Res. 2022 May 15;14(5):3488-3493. eCollection 2022. PMID 35702079
- [Result] Zhou S, Wang L, Chen J, Liu L, Wu X. Effects of individual dietary intervention on blood glucose level and pregnancy outcomes in patients with gestational diabetes mellitus: a retrospective cohort study. Ann Palliat Med. 2021 Sep;10(9):9692-9701. doi: 10.21037/apm-21-2115. PMID 34628895
- [Result] Chen L, Zhang W, Fu A, Zhou L, Zhang S. Effects of WeChat platform-based nursing intervention on disease severity and maternal and infant outcomes of patients with gestational diabetes mellitus. Am J Transl Res. 2022 May 15;14(5):3143-3153. eCollection 2022. PMID 35702129
- [Result] Kapur K, Kapur A, Hod M. Nutrition Management of Gestational Diabetes Mellitus. Ann Nutr Metab. 2021 Feb 1:1-13. doi: 10.1159/000509900. Online ahead of print. PMID 33524988

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT05613920/Prot_SAP_ICF_000.pdf